CLINICAL TRIAL: NCT02045979
Title: Pharmacokinetics and Safety of BI 695501 in Healthy Subjects: a Randomized, Double-blind, Single Dose, Parallel-arm, Active Comparator Clinical Phase I Study
Brief Title: Pharmacokinetics and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1297.8; 2013-003722-84 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 695501

ARMS (3):
- BI 695501 (Experimental): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing BI 695501
  Interventions: Drug: BI 695501
- adalimumab-EU source (Active Comparator): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing adalimumab-EU source
  Interventions: Drug: adalimumab-EU source
- adalimumab-US source (Active Comparator): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing adalimumab-US source
  Interventions: Drug: adalimumab-US source

INTERVENTIONS:
Drug: BI 695501 — BI 695501 single s.c. injection
  Arms: BI 695501
Drug: adalimumab-EU source — adalimumab-EU source single s.c. injection
  Arms: adalimumab-EU source
Drug: adalimumab-US source — adalimumab-US source single s.c. injection.
  Arms: adalimumab-US source

SUMMARY:
Investigate the pharmacokinetics, safety and tolerability of BI695501 and to establish pharmacokinetic similarity of BI 695501 to adalimumab.

ELIGIBILITY:
Inclusion criteria:

Healthy males according to the following criteria:

1. Based upon a complete medical history, including the physical examination, vital signs (blood pressure [BP] and pulse rate [PR]), 12-lead electrocardiogram (ECG), and clinical laboratory tests;
2. Age-greater than or equal to 18 years and less than or equal to 55 years;
3. Body mass index (BMI) =18.5 to =29.9 kg/m2; and
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation.

Exclusion criteria:

1. Any clinically relevant abnormal finding of the medical examination (including blood pressure (BP), pulse rate (PR), and electrocardiogram (ECG) deviating from normal and of clinical relevance;
2. Any evidence of a clinically relevant previous or concomitant disease as judged by the investigator including gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders, or diseases of the central nervous system (such as epilepsy), psychiatric disorders, or neurological disorders;
3. History of relevant orthostatic hypotension, fainting spells, or blackouts;
4. Chronic or relevant acute infections. A negative result for human immunodeficiency virus (HIV), Hepatitis B (Hep B), and hepatitis C (Hep C) is required for participation;
5. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients);
6. Intake of prescribed or over-the-counter drugs with a long half-life (greater than 24 hours) within at least one month or at least 5 half-lives of the respective drug (whichever is longer) prior to administration or during the trial;
7. Previous exposure of a biologic drug;
8. Use of drugs which might reasonably influence the results of the trial prior to dosing and at any time during the trial;
9. Intake of an investigational drug in another trial within two months prior to intake of study medication in this trial or intake of an investigational drug during the course of this trial;
10. Smoker (greater than 10 cigarettes or greater than 3 cigars or greater than 3 pipes/day);
11. Inability to refrain from smoking during days of confinement at the trial site;
12. History of alcohol abuse (estimated average more than 4 units/day);
13. Unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to the study medication administration and until Day 7 post study medication administration;
14. Unwillingness/inability to limit alcohol intake to a maximum of three units per day until e.o.s.;
15. Current drug abuse;
16. Blood donation (more than 100 mL within four weeks prior to administration of the study medication or during the trial);
17. Vigorous exercise 72 hours prior to dosing. Unwilling to avoid vigorous exercise for 7 days post dosing. Contact sport should be avoided during the entire study;
18. Any out-of-range laboratory values considered clinically significant by the investigator; subjects with creatine kinase (CK) values three times the upper limit of normal (ULN) at Day -1 are excluded from participation;
19. Subjects considered unsuitable for inclusion by the investigator (e.g., inability to understand and comply with the study requirements or presence of any condition which, in the opinion of the investigator, would not allow safe participation in the study); or
20. Inability to comply with dietary regimen of trial site.
21. Subjects with known Human immunodeficiency virus (HIV), Acquired Immunodeficiency Syndrome, other clinically significant immunological disorders, or auto-immune disorders, (e.g., Rheumatoid arthritis (RA), lupus erythematosus, scleroderma, etc.);
22. Subject has received a live or attenuated vaccine within 12 weeks prior to enrolling in the trial; or
23. Positive finding in Interferon-gamma-release assay testing (IGRA-T). In cases where at the screening visit the IGRA result is indeterminate, the subject will have a PPD skin test performed, provided that the screening period timeframe can be maintained. If not, the subject will not be enrolled in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2014-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- 1297.8.1001 Boehringer Ingelheim Investigational Site, Antwerp, Belgium
- New Zealand (2):
  - 1297.8.2001 Boehringer Ingelheim Investigational Site, Auckland
  - 1297.8.2002 Boehringer Ingelheim Investigational Site, Christchurch

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Kang J, Eudy-Byrne RJ, Mondick J, Knebel W, Jayadeva G, Liesenfeld KH. Population pharmacokinetics of adalimumab biosimilar adalimumab-adbm and reference product in healthy subjects and patients with rheumatoid arthritis to assess pharmacokinetic similarity. Br J Clin Pharmacol. 2020 Nov;86(11):2274-2285. doi: 10.1111/bcp.14330. Epub 2020 Jun 11. PMID 32363771
- [Derived] Wynne C, Altendorfer M, Sonderegger I, Gheyle L, Ellis-Pegler R, Buschke S, Lang B, Assudani D, Athalye S, Czeloth N. Bioequivalence, safety and immunogenicity of BI 695501, an adalimumab biosimilar candidate, compared with the reference biologic in a randomized, double-blind, active comparator phase I clinical study (VOLTAIRE(R)-PK) in healthy subjects. Expert Opin Investig Drugs. 2016 Dec;25(12):1361-1370. doi: 10.1080/13543784.2016.1255724. PMID 27813422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this trial 324 healthy subjects were randomized into 3 arms.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they (the subject) met all strictly implemented inclusion/exclusion criteria. Subjects were not randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 695501: Subject to receive a single subcutaneous (s.c.) injection from a prefilled syringe containing 40 milligram (mg)/0.8 millilitre (mL) BI 695501 solution.
- US-licensed Humira®: Subject to receive a single subcutaneous (s.c.) injection from a prefilled syringe containing 40 mg/0.8 mL US-licensed Humira®
- EU-approved Humira®: Subject to receive a single subcutaneous (s.c.) injection from a prefilled syringe containing 40 mg/0.8 mL European Union (EU)-approved Humira®.
Period: Overall Study
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Started | 108 (1 subject (not included to the 108) was randomized but did never take any study medication.) | 108 (1 subject (not included to the 108) was randomized but did never take any study medication..) | 108 (1 subject (not included to the 108) was randomized but did never take any study medication.)
Completed | 106 | 107 | 107
Not Completed | 2 | 1 | 1
Not completed — Informed Consent Withdrawn | 2 | 0 | 1
Not completed — not specified above | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all subjects who received the single dose of trial medication.
Groups:
- BI 695501: single s.c. injection 40 mg/0.8 mL BI 695501 solution.
- US-licensed Humira®: single s.c. injection 40 mg/0.8 mL US-licensed Humira®
- EU-approved Humira®: single s.c. injection 40 mg/0.8 mL EU-approved Humira®
- Total: Total of all reporting groups
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira® | Total
Number analyzed (Participants) | 108 | 108 | 108 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (11) | 31 (11) | 30 (12) | 31 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 108 | 108 | 108 | 324

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve (AUC) From Time Zero to Infinity (AUC 0-∞) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to infinity (AUC 0-∞) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  Abbreviation used: Pharmacokinetics (PK).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312, 480, 648, 1032, 1320 h post dosing and on day 71 post dosing.
Population: PK analysis set consisted of all randomized subjects who received the single dose of trial medication (BI 695501, US-licensed - or EU-approved Humira®), had at least one evaluable primary PK endpoint and were without important protocol deviations or violations thought to significantly affect the PK of BI 695501, US-licensed - or EU-approved Humira®
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)*hour (h)/millilitre (mL)
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 106 | 105 | 105
microgram (µg)*hour (h)/millilitre (mL) | 2630 (52.4) | 2470 (51.2) | 2650 (38.5)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — PK similarity of the two treatments was to be concluded if the 90% CI for the ratio of adjusted geometric means was within 80.00 - 125.00 percent (%); ratio of the geometric means = 108.62, 90% CI 2-sided [98.50 to 119.79] — An analysis of covariance (ANCOVA) model on the logarithmic scale with fixed effects for treatment and trial site as well as age (as recorded at the time of informed consent) and body weight (as recorded at baseline) as continuous covariates
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — PK similarity of the two treatments was to be concluded if the 90% CI for the ratio of adjusted geometric means was within 80.00 - 125.00 %; ratio of the geometric means = 101.27, 90% CI 2-sided [92.45 to 110.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 94.02, 90% CI 2-sided [86.01 to 102.78] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC0-tz) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve from time zero to last measurable concentration (AUC0-tz) of BI 695501, US-licensed Humira® or EU-approved Humira®.
Time Frame: as for outcome 1
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 106 | 107 | 106
µg*h/mL | 2440 (47.8) | 2300 (45.1) | 2480 (33.5)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 107.32, 90% CI 2-sided [98.49 to 116.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 99.93, 90% CI 2-sided [92.15 to 108.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 93.66, 90% CI 2-sided [86.76 to 101.11] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Concentration (Cmax) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Maximum concentration (Cmax) of BI 695501, US-licensed Humira® or EU-approved Humira®.
Time Frame: as for outcome 1
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 108 | 107
µg/mL | 3.907 (34.1) | 3.900 (34.5) | 4.140 (30.4)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 100.85, 90% CI 2-sided [95.15 to 106.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 96.39, 90% CI 2-sided [91.06 to 102.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ratio of the geometric means = 95.93, 90% CI 2-sided [90.83 to 101.33] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUC (0-168) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to 168 hours post dose (AUC 0-168) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  PK is the abbreviation for Pharmacokinetic(s).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168 hours post dosing
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 108 | 107
µg*h/mL | 480 (41.1) | 493 (40.7) | 513 (39.9)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% Confidence Interval (CI) for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 98.30, 90% CI 2-sided [91.54 to 105.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 96.05, 90% CI 2-sided [89.27 to 103.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 98.11, 90% CI 2-sided [91.42 to 105.27] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: AUC (0-312) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to 312 hours post dose (AUC 0-312) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  PK is the abbreviation for Pharmacokinetic(s).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312 hours post dosing
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 108 | 107
µg*h/mL | 957 (36.5) | 967 (34.9) | 1010 (31.6)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 99.61, 90% CI 2-sided [93.66 to 105.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 97.19, 90% CI 2-sided [91.39 to 103.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 97.97, 90% CI 2-sided [92.58 to 103.68] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC (0-480) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to 480 hours post dose (AUC 0-480) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  PK is the abbreviation for Pharmacokinetic(s).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312, 480 hours post dosing
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 108 | 107
µg*h/mL | 1400 (35.8) | 1390 (32.2) | 1440 (28.0)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 101.23, 90% CI 2-sided [95.45 to 107.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 98.83, 90% CI 2-sided [93.27 to 104.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 98.01, 90% CI 2-sided [93.15 to 103.11] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: AUC (0-648) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to 648 hours post dose (AUC 0-648) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  PK is the abbreviation for Pharmacokinetic(s).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312, 480, 648 hours post dosing
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 108 | 107
µg*h/mL | 1730 (37.0) | 1680 (33.2) | 1760 (27.2)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 103.68, 90% CI 2-sided [97.47 to 110.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 100.16, 90% CI 2-sided [94.37 to 106.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 97.02, 90% CI 2-sided [92.07 to 102.24] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: AUC (0-1032) of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to 1032 hours post dose (AUC 0-1032) of BI 695501, US-licensed Humira® or EU-approved Humira® PK is the abbreviation for Pharmacokinetic(s).
Time Frame: at -1 hour (h) (pre dosing) and 1h, 4, 8, 12, 24, 48, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312, 480, 648, 1032 hours post dosing
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 107 | 106 | 106
µg*h/mL | 2190 (41.4) | 2080 (38.5) | 2210 (29.1)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 106.57, 90% CI 2-sided [99.07 to 114.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 100.94, 90% CI 2-sided [94.24 to 108.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 95.37, 90% CI 2-sided [89.53 to 101.60] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: AUC 0-∞,Obs of BI 695501, US-licensed Humira® or EU-approved Humira®
Description: Area under the concentration time curve (AUC) from time zero to infinity (AUC 0-∞) based on the last observed concentration at time of last measureable concentration (tz) of BI 695501, US-licensed Humira® or EU-approved Humira®.
  PK is the abbreviation of Pharmacokinetic(s).
Time Frame: as for outcome 1
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 106 | 105 | 105
µg*h/mL | 2630 (52.6) | 2470 (51.3) | 2640 (38.5)
Statistical Analysis 1: Comparison: BI 695501 vs US-licensed Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 108.70, 90% CI 2-sided [98.54 to 119.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 101.36, 90% CI 2-sided [92.51 to 111.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: US-licensed Humira® vs EU-approved Humira®; Test type: Non-Inferiority or Equivalence — No formal testing; two-sided 90% CI for the ratio of adjusted geometric means was calculated; ratio of the geometric means = 94.04, 90% CI 2-sided [86.01 to 102.82] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number (Proportion) of Subjects With Drug Related Adverse Events
Description: All events with an onset after the first administration of the trial medication up to a period of 70 days after the last administration of the trial medication (i.e., end of the REP) was assigned to the treatment phase for evaluation and was defined as a treatment-emergent AE (TEAE). A treatment-related AE was defined as any TEAE assessed by the investigator as related to the trial medication.
  All safety data were displayed and analyzed using descriptive statistical methods. No formal inferential analyses were planned for safety comparisons. Tabulations of frequencies and proportions, as appropriate were used for the evaluation of categorical (qualitative) data, and tabulations of descriptive statistics were used to analyze continuous (quantitative) data.
Time Frame: Day 1 through Day 71
Population: The safety analysis set consisted of all subjects who received the single dose of trial medication (BI 695501, US-licensed Humira® or EU-approved Humira®).
Measure: Number; unit: participants
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Number analyzed (Participants) | 108 | 108 | 108
participants | 21 | 29 | 28

ADVERSE EVENTS:
Time Frame: Day 1 (first administration of trial medication) until day 71
Arm/Group | BI 695501 | US-licensed Humira® | EU-approved Humira®
Serious Adverse Events (participants affected / at risk) | 3/108 | 3/108 | 2/108
Other Adverse Events (participants affected / at risk) | 51/108 | 52/108 | 51/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=108) | US-licensed Humira® (N=108) | EU-approved Humira® (N=108)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=108) | US-licensed Humira® (N=108) | EU-approved Humira® (N=108)
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 7 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 19 | 17 | 22
Headache (Nervous system disorders) | 25 | 25 | 28
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.